CLINICAL TRIAL: NCT04448626
Title: Micro-environment Involvement in Muscle Alteration Induced by Copd Exacerbation
Brief Title: Micro-environment Involvement in Muscle Alteration Induced
Acronym: MicAMI-BPCO
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: APARD Fonds de dotation (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0137
Record Dates: First submitted 2020-06-15; First posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Exacerbations; Skeletal Muscle Atrophy
Keywords: COPD Exacerbation; Muscle atrophy; Inflammation; Oxidative stress; Biomarkers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Muscular Atrophy; Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy subject: Healthy subject
- Stable COPD patients: Stable COPD patients
- Exacerbation COPD patients: Exacerbation COPD patients

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is characterized by persistent airway obstruction and inflammatory response of the lungs and bronchi. Episodes of exacerbations contribute to increase the severity and prognosis of the disease. Muscle dysfunction (loss of strengh and muscle mass) is one of comorbidities affecting 30% to 60% of patients and playing a key role in their prognosis. During exacerbation, some studies have suggested an association between muscle dysfunction and modifications of inflammatory circulating factors such as CRP, TNF-alpha, IL- 6, IL8, but no exhaustive study has identified precisely one (or more) biomarker(s) that can induce this muscle wasting during the exacerbation of COPD. Our hypothesis is that the serum of exacerbated COPD patients represents a deleterious microenvironment for the muscle cells which would amplify the mechanisms of atrophy linked to hospitalization. Our team has already developed a cell culture model to study the effects of the plasma microenvironment on atrophy of cultured myotubes. The investigators have shown that the serum of COPD patients can induce muscle atrophy.

The objectives of this study are : 1/ to evaluate the effects of circulating pro-inflammatory factors on atrophy and the myogenic capacities of muscle cells; and 2/ to identify one (or more) circulating biomarker (s) that may be responsible for the muscle damage induced by the microenvironment of hospitalized patients for exacerbation of COPD. First, myotubes and myoblasts of healthy subjects will be cultivated with 9 exacerbation copd patient serum or 9 copd patient serum or 9 healthy subject serum. Myotube diameters, atrophy, inflammatory and oxidative stress markers and alteration of the myogenic capacity of satellite cells will be compared between three groups. Second, the differential expression of circulating proinflammatory molecules will be compared in the serum of the three groups. Identifying circulating factors associated with muscle weakness is a necessary step to better understand the mechanisms and consider a personalized therapeutic approach that can improve the functional and clinical prognosis of disease.

.

ELIGIBILITY:
Inclusion criteria 1/ for COPD patients hospitalized for exacerbation:

* Hospitalization for COPD exacerbation 2/ for COPD patients
* COPD patients GOLD II à IV
* Not having followed respiratory réhabilitation stay for at least one year 3/ for Healthy subjects
* healthy and sedentary (Voorips score <9)

Exclusion criteria:

1. for COPD patients hospitalized for exacerbation:

   * concomitant acute cardiac évent
   * trachéal intubation with mechanical ventilation
   * chronic respiratory disease other than COPD
   * locomotor, neurologic or psychiatric comorbidities
2. for COPD patients

   * Exacerbation with récent hospitalization (<4 weeks)
   * Neurologic comorbidity
3. for Healthy subjects - long term drug treatment with proven central effects

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COPD patients hospitalized for exacerbation in Montpellier university hospital, France.
  COPD patients recruited in Clinique du Souffle, La Vallonie, Lodève, France. Healthy volunteer subject recruited in Clinique du Souffle, La Vallonie, Lodève, France.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Effects evaluation of circulating pro-inflammatory factors on atrophy | 6 months
  Atrophy marker evaluation in cultured muscle cells (myotubes)
  * cultured myotube diameter exposed to the three serum groups (immunofluorescence)
  * atrophy (ubiquitin proteasome system, proteolytic autophagy pathway), inflammatory (TNF-alpha, IL-6, IL-8…) and oxidative stress (ROS, lipid peroxidation) markers expressed by cells exposed to the three serum groups (PCR et WesternBlot)
Effects evaluation of circulating pro-inflammatory factors on the myogenic capacities of muscle cells | 6 months
  Myogenic capacities of cultured muscle cells (myoblastes)
  * inflammatory (TNF-alpha, IL-6, IL-8…) and oxidative stress (ROS, lipid peroxidation) markers expressed by cells exposed to the three serum groups (PCR et WesternBlot)
  * regeneration markers (Notch and myogenesis signaling pathways) expressed by cells exposed to the three serum groups (PCR et WesternBlot)

SECONDARY OUTCOMES:
Identification of one (or more) circulating biomarker (s) | 3 months
  Identification of one (or more) circulating biomarker (s) that may be responsible for the muscle alteration induced by the microenvironment of patient in exacerbation of COPD

CONTACTS AND LOCATIONS:
Overall Officials: Maurice HAYOT, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Background] Spruit MA, Gosselink R, Troosters T, Kasran A, Gayan-Ramirez G, Bogaerts P, Bouillon R, Decramer M. Muscle force during an acute exacerbation in hospitalised patients with COPD and its relationship with CXCL8 and IGF-I. Thorax. 2003 Sep;58(9):752-6. doi: 10.1136/thorax.58.9.752. PMID 12947130
- [Background] Crul T, Testelmans D, Spruit MA, Troosters T, Gosselink R, Geeraerts I, Decramer M, Gayan-Ramirez G. Gene expression profiling in vastus lateralis muscle during an acute exacerbation of COPD. Cell Physiol Biochem. 2010;25(4-5):491-500. doi: 10.1159/000303054. Epub 2010 Mar 23. PMID 20332630
- [Background] Crul T, Spruit MA, Gayan-Ramirez G, Quarck R, Gosselink R, Troosters T, Pitta F, Decramer M. Markers of inflammation and disuse in vastus lateralis of chronic obstructive pulmonary disease patients. Eur J Clin Invest. 2007 Nov;37(11):897-904. doi: 10.1111/j.1365-2362.2007.01867.x. Epub 2007 Sep 20. PMID 17883420
- [Background] Catteau M, Gouzi F, Blervaque L, Passerieux E, Blaquiere M, Ayoub B, Bughin F, Mercier J, Hayot M, Pomies P. Effects of a human microenvironment on the differentiation of human myoblasts. Biochem Biophys Res Commun. 2020 May 14;525(4):968-973. doi: 10.1016/j.bbrc.2020.03.020. Epub 2020 Mar 12. PMID 32173533